CLINICAL TRIAL: NCT02892604
Title: Pilot Evaluation Study of the Feasibility of a Permanent Use in Free-life of inControl Artificial Pancreas System for the Treatment of Type 1 Diabetes
Brief Title: Study the Feasibility of Permanent Use of inControl for the Treatment of Type 1 Diabetes
Acronym: IDCLTraining
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough participants
Sponsor: University Hospital, Montpellier (Other)
Collaborators: MEDBIOMED, Montpellier, France (Unknown); Jaeb Center for Health Research (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9722
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; artificial pancreas; closed-loop insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- insulin delivery driven by inControl (Experimental): Closed-loop insulin delivery using inControl AP system is assessed for two weeks, 24/7.
  Connection of continuous glucose monitoring (CGM) system and insulin pump to inControl AP platform, all wireless and wearable, in free-life conditions Insulin from the pump is delivered according to the closed-loop algorithm fed by CGM data.
  Interventions: Device: insulin pump to inControl AP platform

INTERVENTIONS:
Device: insulin pump to inControl AP platform — Insulin from the pump is delivered according to the closed-loop algorithm fed by CGM data.

SUMMARY:
A new version of the DiAs artificial pancreas (AP) system has been developed in view of wide scale outpatient trials. Denominated as inControl , it includes improved user interface and communication modules while closed-loop algorithms remain similar. During this pilot study, the investigators will evaluate this new version of AP for a two-week period during which the patients will use it for closed-loop insulin delivery 24/7 The main goal is train the clinical team with the new system and collect patient opinions on system acceptance from questionnaires. If this trial is conclusive, a randomized 6-month multicentre study including 240 patients will be initiated. A total of 5 patients will be included in this training study over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus since more than one year, treated by insulin since at least one year
* Treatment by insulin pump since at least 6 months
* Glycated hemoglobin (HbA1c) below 10.5% at inclusion visit
* For women of child bearing age, no current pregnancy and use of an efficient contraception during the whole research participation
* Agreement on no use of drugs or products used for reduction of blood glucose levels, such as metformin or GLP1 analogs, except if this therapy has been used for at least 3 months before study start
* Agreement on stopping closed-loop insulin delivery after acetaminophen use and 4 following hours
* Agreement on suspending use of patient CGM device during the study period while study CGM will be used
* Access to the internet and a mobile phone network at home
* Agreement on following study procedures
* Affiliation to the French social security system or a similar healthcare coverage system
* Mandatory written informed consent

Exclusion Criteria:

* Need for chronic use of acetaminophen
* Start of use of drugs or products used for reduction of blood glucose levels, such as metformin or GLP1 analogs during the 3 months before inclusion
* Hemophilia or other coagulation disorders
* Psychological and/or cognitive troubles which may impair the appropriate following of study procedures
* Diabetic ketoacidosis during the last 6 months
* Acute cardiovascular event during the last 12 months
* Severe hypoglycaemia with convulsions or loss of conscience during the last 12 months
* Use of a therapy with significant impact on glucose metabolism
* Cystic fibrosis
* Lack of nearby third-party assistance availability in case of troubles
* Malignant disease, except if considered as cured since at least 10 years
* Impaired kidney function (serum creatinin > 150 umol/L)
* Impaired liver status (ALAT or ASAT > 2-times upper normal limit)
* Active gastroparesis
* Acute adrenocortical event
* Alcohol or narcotics abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-24 (Actual)

PRIMARY OUTCOMES:
Percent time of active insulin closed-loop delivery | 2 weeks
  Percent time while AP system is active permanently

SECONDARY OUTCOMES:
Percent time with blood glucose in target range | 2 weeks
  Percent time while blood glucose is kept in safe 70-180 mg/dl range

CONTACTS AND LOCATIONS:
Overall Officials: Eric M RENARD, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided